CLINICAL TRIAL: NCT01319357
Title: Effects of Saxagliptin on Endothelial Function in Patients With Type 2 Diabetes
Brief Title: Effects of Saxagliptin on Endothelial Function
Acronym: ESENDI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Roland E. Schmieder, Prof. Dr. med., University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SAXA24011980GLIPTIN
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Saxagliptin (Active Comparator): saxagliptin 5 mg/day during 6 weeks
  Interventions: Drug: Saxagliptin

INTERVENTIONS:
Drug: Saxagliptin — orally 5 mg/d for 6 weeks
  Other Names: Onglyza
  Arms: Saxagliptin
Drug: Placebo — orally for 6 weeks
  Arms: Placebo

SUMMARY:
Diabetes mellitus is a metabolic disease with a growing prevalence worldwide. Currently available therapies for type 2 diabetes have various limitations and are associated with increased risk of hypoglycemia, weight gain, gastrointestinal side effects or edema and heart failure.

A new and promising class of drugs are the gliptins. Several efficacy studies demonstrated a significant improvement of HbA1c with gliptins. In addition, gliptins improved fasting as well as prandial glucose levels and did not induce weight gain. Due to these positive metabolic effects in combination with a very small spectrum of side effects gliptins might very well be part of the standard therapy for type 2 diabetes in the future.

Apart form surrogate parameters like reduction of fasting and postprandial blood glucose levels or improvement of HbA1c, the effect of gliptins on micro- and macrovascular function and cardiovascular outcome has not been the primary focus of current studies. Diabetes mellitus is strongly associated with microangiopathy and macroangiopathy and is a strong independent risk factor for cardiovascular disease and cardiovascular mortality. Endothelial dysfunction which plays a crucial role in the atherosclerotic process is commonly observed in patients with diabetes mellitus and already prediabetes and has - amongst other factors - been linked to fasting and postprandial hyperglycemia. Taken into account that gliptins reduce hyperglycemia and hyperglycemic peaks by preventing inactivation of GLP-1, which exerted beneficial effects on the endothelium in previous studies it is of major interest whether therapy with gliptins improves endothelial function.

DETAILED DESCRIPTION:
Diabetes mellitus is a metabolic disease with a growing prevalence worldwide, affecting 171 million people in 2000 and an expected 366 million people in 2030 [1].. Currently available therapies for type 2 diabetes have various limitations and are associated with increased risk of hypoglycemia, weight gain, gastrointestinal side effects or edema and heart failure.

A new and promising class of drugs are the gliptins. Gliptins act by inhibiting the enzyme dipeptidyl peptidase-4 (DPP-4), which is responsible for the rapid inactivation of glucagon-like peptide-1 (GLP-1) - an incretin hormone of the gut [2-4], thereby enhancing and prolonging the effects of GLP-1. GLP-1 - member of the incretin hormones - is released into the blood after meal ingestion and stimulates the insulin secretion in a glucose dependent manner. This accounts for the marked prandial insulin response, which prevents prandial hyperglycemia. Several efficacy studies demonstrated a significant improvement of HbA1c with gliptins. In addition, gliptins improved fasting as well as prandial glucose levels and did not induce weight gain. Due to these positive metabolic effects in combination with a very small spectrum of side effects gliptins might very well be part of the standard therapy for type 2 diabetes in the future.

Apart form surrogate parameters like reduction of fasting and postprandial blood glucose levels or improvement of HbA1c, the effect of gliptins on micro- and macrovascular function and cardiovascular outcome has not been the primary focus of current studies. However, infusion of GLP-1, the incretin hormone affected by gliptins has been reported to ameliorate endothelial dysfunction in patients suffering from coronary artery disease [5] and it was recently shown that infusion of GLP-1 into healthy human subjects increases both normal and ACh-induced vasodilatation [6]. In studies on rats with diabetes, GLP-1 infusion nearly re-established their normal vascular tone [7] and there are further data from experimental animals that indicate a beneficial effect of GLP-1 on endothelial function [8].

Diabetes mellitus is strongly associated with microangiopathy and macroangiopathy and is a strong independent risk factor for cardiovascular disease and cardiovascular mortality [9]. Endothelial dysfunction which plays a crucial role in the atherosclerotic process is commonly observed in patients with diabetes mellitus and already prediabetes and has - amongst other factors - been linked to fasting and postprandial hyperglycemia. Taken into account that gliptins reduce hyperglycemia and hyperglycemic peaks by preventing inactivation of GLP-1, which exerted beneficial effects on the endothelium in previous studies it is of major interest whether therapy with gliptins improves endothelial function of the micro- and macrovasculature and thereby might prove to affect cardiovascular morbidity and mortality in diabetic patients in the long term. The retina offers the unique opportunity to directly visualize and investigate the microvasculature in vivo [10-14].

References

1. Wild S, Roglic G, Green A, Sicree R, King H: Global prevalence of diabetes: Estimates for the year 2000 and projections for 2030. Diabetes Care 2004;27:1047-1053.
2. Deacon CF, Ahren B, Holst JJ: Inhibitors of dipeptidyl peptidase iv: A novel approach for the prevention and treatment of type 2 diabetes? Expert Opin Investig Drugs 2004;13:1091-1102.
3. Deacon CF: Therapeutic strategies based on glucagon-like peptide 1. Diabetes 2004;53:2181-2189.
4. Holst JJ, Deacon CF: Glucagon-like peptide-1 mediates the therapeutic actions of dpp-iv inhibitors. Diabetologia 2005;48:612-615.
5. Nystrom T, Gutniak MK, Zhang Q, Zhang F, Holst JJ, Ahren B, Sjoholm A: Effects of glucagon-like peptide-1 on endothelial function in type 2 diabetes patients with stable coronary artery disease. Am J Physiol Endocrinol Metab 2004;287:E1209-1215.
6. Basu A, Charkoudian N, Schrage W, Rizza RA, Basu R, Joyner MJ: Beneficial effects of glp-1 on endothelial function in humans: Dampening by glyburide but not by glimepiride. Am J Physiol Endocrinol Metab 2007;293:E1289-1295.
7. Ozyazgan S, Kutluata N, Afsar S, Ozdas SB, Akkan AG: Effect of glucagon-like peptide-1(7-36) and exendin-4 on the vascular reactivity in streptozotocin/nicotinamide-induced diabetic rats. Pharmacology 2005;74:119-126.
8. Yu M, Moreno C, Hoagland KM, Dahly A, Ditter K, Mistry M, Roman RJ: Antihypertensive effect of glucagon-like peptide 1 in dahl salt-sensitive rats. J Hypertens 2003;21:1125-1135.
9. Laakso M: Hyperglycemia and cardiovascular disease in type 2 diabetes. Diabetes 1999;48:937-942.
10. Delles C, Michelson G, Harazny J, Oehmer S, Hilgers KF, Schmieder RE: Impaired endothelial function of the retinal vasculature in hypertensive patients. Stroke 2004;35:1289-1293.
11. Harazny JM, Ritt M, Baleanu D, Ott C, Heckmann J, Schlaich MP, Michelson G, Schmieder RE: Increased wall:Lumen ratio of retinal arterioles in male patients with a history of a cerebrovascular event. Hypertension 2007;50:623-629.
12. Ritt M, Schmieder RE: Wall-to-lumen ratio of retinal arterioles as a tool to assess vascular changes. Hypertension 2009;54:384-387.
13. Oehmer S, Harazny J, Delles C, Schwarz T, Handrock R, Michelson G, Schmieder RE: Valsartan and retinal endothelial function in elderly hypertensive patients. Blood Press 2006;15:185-191.
14. Ott C, Schlaich MP, Harazny J, Schmidt BM, Michelson G, Schmieder RE: Effects of angiotensin ii type 1-receptor blockade on retinal endothelial function. J Hypertens 2008;26:516-522.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes mellitus defined by fasting glucose ≥126 mg/dl or HbA1c ≥6.5% or on blood glucose lowering medication
* Age of 18 - 75 years
* Male and Female patients are eligible. Females of child bearing potential or within two years of the menopause are only eligible if pregnancy test at the screening visit is negative and they use adequate contraceptive precautions during the trial.
* The patient must demonstrate that she/he is able and willing to perform blood glucose measurements as necessary for Home Blood Glucose Monitoring by herself/himself after it was demonstrated to her/him.

Exclusion Criteria:

* Any other form of diabetes mellitus than type 2 diabetes mellitus
* Patients with more than on one blood glucose lowering medication or on insulin therapy
* Last measured HbA1c > 11%
* Blood pressure levels ≥180/110 mmHg
* Body mass index >50 kg/m²
* Triglyceride levels >1000 mg/dl
* HDL-cholesterol levels <25 mg/dl
* Estimated creatinine clearance < 50 ml/min/1.73m²
* Macroalbuminuria defined by urinary albumine-to-creatinine ratio > 300 mg/g
* Known liver function test >3 times upper limit of normal
* Pregnant or breast-feeding patients
* Current or previous (within 6 months) treatment with an incretin-based therapy such as DPP 4 inhibitors and/or GLP-1 mimetics
* Any patient currently receiving chronic (>30 consecutive days) treatment with an oral corticosteroid
* Acute cardiovascular event (including myocardial infarction, unstable angina pectoris, percutaneous coronary intervention, heart failure, stroke, TIA. PRIND, intracerebral bleeding) <6 months prior to screening visit (visit 1)
* Diabetic retinopathy
* History of epilepsia or history of seizures
* Patients being treated for severe auto immune disease e.g. lupus
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca and BMS or representative staff and/or staff at the study site)
* Previous randomisation in the present study
* Participation in another clinical study within 30 days prior to visit 1
* Individuals at risk for poor protocol or medication compliance
* Subject who do not give written consent, that pseudonymous data will be transferred in line with the duty of documentation and the duty of notification according to § 12 and § 13 GCP-V

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
effect of saxagliptin compared to placebo on endothelial and vascular function of the retinal circulation | after 6 weeks of treatment with saxagliptin vs. 6 weeks of treatment with placebo (12 weeks in all)
  retinal circulation. By applying Scanning-Laser-Doppler-Flowmetry, the change of retinal capillary flow after i.v. L-NMMA application

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, MD, Principal Investigator — University of Erlangen-Nürnberg
Locations (1):
- Clinical Research Center, Department of Nephrology and Hypertension, University of Erlangen-Nuremberg, Erlangen, Germany

REFERENCES:
- [Result] Ott C, Raff U, Schmidt S, Kistner I, Friedrich S, Bramlage P, Harazny JM, Schmieder RE. Effects of saxagliptin on early microvascular changes in patients with type 2 diabetes. Cardiovasc Diabetol. 2014 Jan 14;13:19. doi: 10.1186/1475-2840-13-19. PMID 24423149
- [Derived] Staef M, Ott C, Kannenkeril D, Striepe K, Schiffer M, Schmieder RE, Bosch A. Determinants of arterial stiffness in patients with type 2 diabetes mellitus: a cross sectional analysis. Sci Rep. 2023 Jun 2;13(1):8944. doi: 10.1038/s41598-023-35589-4. PMID 37268640
- [Derived] Kannenkeril D, Bosch A, Harazny J, Karg M, Jung S, Ott C, Schmieder RE. Early vascular parameters in the micro- and macrocirculation in type 2 diabetes. Cardiovasc Diabetol. 2018 Sep 19;17(1):128. doi: 10.1186/s12933-018-0770-4. PMID 30231923